CLINICAL TRIAL: NCT00341523
Title: Early Detection of Esophageal Cancer
Status: Terminated | Type: Observational
Why Stopped: Administratively closed by the IRBO
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 999995026; OH95-C-N026; NCT00005885 (obsolete NCT alias)
Record Dates: First submitted 2006-06-19; First posted 2006-06-21 (Estimated); Last update posted 2024-05-01 (Actual); Status verified 2024-04

CONDITIONS: Esophageal Neoplasms; Stomach Neoplasms; Endoscopy, Gastrointestinal; Digestive System Endoscopic Surgical Procedures; Cytology
Keywords: Cytology; Endoscopy; Esophageal Cancer; Early Detection; Treatment; Natural History
MeSH Terms: conditions — Esophageal Neoplasms; Stomach Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- 1: Chinese adults at high risk for esophageal cancer

SUMMARY:
Esophageal cancer is a common malignancy with a very poor prognosis. The principal reason for its poor prognosis is that most tumors are asymptomatic and go undetected until they have spread beyond the esophageal wall and are unresectable. Significant reduction in esophageal cancer mortality will require successful strategies to diagnose and treat more cases at earlier, more curable stages of disease. A successful early detection program will require an accurate, patient-acceptable screening test, confirmatory tests that can localize precursor and early invasive lesions, and one or more curative therapies that are acceptable to asymptomatic patients. This project includes five studies designed to evaluate techniques that may be useful in such an early detection program:

1. The Cytology Sampling Study will estimate and compare the sensitivity of several cytologic samplers for identifying biopsy-proven dysplasia and cancer of the esophagus.
2. The Mucosal Staining Study will evaluate whether mucosal straining can improve endoscopic localization of esophageal dysplasia and cancer.
3. The Endoscopic Staging Study will evaluate how accurately endoscopic techniques can stage dysplasia and early invasive cancer of the esophagus.
4. The Endoscopic Therapy Pilot Study will evaluate the feasibility, safety, acceptability and preliminary efficacy of endoscopic therapies for removing or ablating focal high-grade dysplasias and early invasive cancers of the esphagus.
5. The Chemoregression Study will evaluate the ability of oral chemopreventive agents to reduce progression or cause regression of low-grade squamous dysplasia of the esophagus.

This project will be carried out in Linxian, China, a county with extraordinary rates of esophageal cancer and a correspondingly high prevalence of the asymptomatic precursor and early invasive lesions that are needed for these studies. The project will be a collaborative effort of investigators from NCI, the Cancer Institute of the Chinese Academy of Medical Sciences, and several U.S. universities.

DETAILED DESCRIPTION:
Esophageal squamous cell carcinoma (ESCC) is a major cause of death in the central

Asian esophageal cancer belt and human papillomavirus (HPV) has been proposed as a potential cause. While several HPV-associated cancers have been identified (e.g., cervical, tonsillar), the role of HPV in esophageal carcinogenesis remains unclear. Estimates of the prevalence of HPV in ESCC in Henan province, which lies in the central Asian esophageal cancer belt and of which Linxian is a part, have varied from 0-78%. Contamination of specimens may contribute to this variation, as may differences in HPV detection techniques. With the imminent availability of an effective HPV vaccine, it is critical to determine if HPV is or is not involved in ESCC in Linxian given the potential for cancer prevention through use of the

vaccine if HPV is involved. OBJECTIVES: The overall objective is to test the hypothesis that HPV is involved in the pathogenesis of ESCC in Linxian, China.

We will 1) determine the prevalence of HPV DNA in ESCC tumors and 2) evaluate the activity of HPV in HPV DNA-positive cases.

ELIGIBILITY:

This study will be conducted among adult patients with ESCC presenting for esophagectomy at Yaocun Commune Hospital in Linxian, China.

DESIGN: This case series study will collect demographic and clinical data from medical records and will use rigorous sterile procedures to obtain biologic specimens (blood, tumor, nontumor) from patients with ESCC. The presence of HPV DNA in tumor specimens will be evaluated using PCR with L1, E6, and E7-based primers. The activity of HPV in HPV DNA-positive cases will be assessed by immunohistochemistry for p16 (ink4a) over-expression, RT-PCR for E6/E7 mRNA expression, and amplification of papillomavirus oncogene transcripts (APOT) for HPV integration in tumor specimens. Nontumor specimens will also be examined for the presence of HPV DNA, and serum will be tested for HPV 16 and HPV 18 E6/E7 seropositivity as a marker of HPV-associated cancer.

ELIGIBILITY:
* INCLUSION CRITERIA:

Resident of Linxian, Henan Province, People's Republic of China.

40-69 years of age at the time of EGD screening.

Visible esophageal lesions with mild or moderate squamous dysplasia found at the t(-6) EGD screening exam.

Confirmation of a visible index lesion at the t(0)EGD baseline exam.

Willing to abstain from chronic NSAID use (defined as greater than 3 times per week for more than 2 weeks), with the exception of low-dose aspirin (less than or equal to 100 mg per day), for the duration of the study.

If a subject is female and of child-bearing potential (premenopausal or less than 2 years postmenopausal and not surgically sterile), she must be willing to use adequate contraception (abstinence, IUD, birth control pills, or spermicidal gel with diaphragm or condom) for the duration of the study.

Appropriate laboratory values within 2 weeks of the baseline evaluation for:

hemoglobin greater than 11.0 g/dl;

WBC greater than 3000/mm(3);

platelet count greater than 100,000;

creatinine less than or equal to 1.5 times the upper limit of normal;

AST less than or equal to 1.5 times the upper limit of normal;

Alkaline phosphatase less than or equal to 1.5 the upper limit of normal;

Pregnancy test negative serum or urine (women of childbearing potential only).

Only those patients with mild or moderate dysplasia based on the t(-6) histology and endoscopically visible lesions at the t(0) evaluation will be eligible for participation and inclusion in the study.

To be eligible at t(0), subjects must have a confirmed, endoscopically visible lesion.

EXCLUSION CRITERIA:

Diagnosed cancer at any site, except non-melanoma skin cancer.

Current symptoms suggestive of an upper gastrointestinal tract malignancy, including dysphagia, odynophagia, hematemesis, or weight loss of greater than 10% body weight within the past 6 months.

Contraindications to the EGD exams, including hypersensitivity to lidocaine or iodine, uncontrolled congestive heart failure, unstable angina, bleeding disorder or severe pulmonary disease.

Contraindications to use of the intervention agents, including hypersensitivity to selenomethionine, COX-2 inhibitors, NSAIDs, salicylates, or sulfonamides.

Treated for peptic ulcer disease within the past month prior to the baseline evaluation.

Acute or chronic kidney disease, liver disease, or asthma.

Pregnant or nursing an infant.

Other serious health condition that might preclude study completion (at the discretion of the investigators).

Currently using fluconazole or lithium.

Ages: 21 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Chinese adults at high risk for esophageal cancer, and Chinese adults presenting with esophageal cancer in Linxian, China
Sampling Method: Non-Probability Sample
Enrollment: 6864 (Actual)
Dates: Start 2016-11-01 (Actual); Primary Completion 2024-04-29 (Actual); Study Completion 2024-04-29 (Actual)

PRIMARY OUTCOMES:
esophageal squamous dysplasia and cancer | single time point when samples are collected
  These case series studies have collected demographic and clinical data from medical records and patient questionnaires and have collected biological samples.

SECONDARY OUTCOMES:
Esophageal squamous cell carcinoma (ESCC) | Clinical diagnosis of ESCC
Death from any cause | Death

CONTACTS AND LOCATIONS:
Overall Officials: Christian Abnet, Ph.D., Principal Investigator — National Cancer Institute (NCI)
Locations (1):
- Cancer Institute and Hospital, Chinese Academy of Medical Sciences, Beijing, China

REFERENCES:
- [Background] Pan QJ, Roth MJ, Guo HQ, Kochman ML, Wang GQ, Henry M, Wei WQ, Giffen CA, Lu N, Abnet CC, Hao CQ, Taylor PR, Qiao YL, Dawsey SM. Cytologic detection of esophageal squamous cell carcinoma and its precursor lesions using balloon samplers and liquid-based cytology in asymptomatic adults in Llinxian, China. Acta Cytol. 2008 Jan-Feb;52(1):14-23. doi: 10.1159/000325430. PMID 18323271
- [Background] Dawsey SM, Fleischer DE, Wang GQ, Zhou B, Kidwell JA, Lu N, Lewin KJ, Roth MJ, Tio TL, Taylor PR. Mucosal iodine staining improves endoscopic visualization of squamous dysplasia and squamous cell carcinoma of the esophagus in Linxian, China. Cancer. 1998 Jul 15;83(2):220-31. PMID 9669803
- [Background] Taylor PR, Abnet CC, Dawsey SM. Squamous dysplasia--the precursor lesion for esophageal squamous cell carcinoma. Cancer Epidemiol Biomarkers Prev. 2013 Apr;22(4):540-52. doi: 10.1158/1055-9965.EPI-12-1347. PMID 23549398